CLINICAL TRIAL: NCT03086291
Title: A Phase I Study of High Dose Simvastatin in Patients With Gastrointestinal Tract Cancer Who Failed to Standard Chemotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-02-138
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Simvastatin 5-10mg/kg bid for 7 days and 14 days off treatment for 21 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- simvastatin (Experimental): One arm Simvastatin 5-10mg/kg bid for 7 days and 14 days off treatment for 21 days Cohort 1: 7.5 mg/kg bid for 7 days 14 days off Cohort 2: 10 mg/kg bid for 7 days 14 days off Cohort 3: ( ) mg/kg bid for 7 days 14 days off (to be determined based on PK data of cohort 1 and 2) Q 3 weeks
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 5-10mg/kg bid for 7 days and 14 days off treatment for 21 days

SUMMARY:
Simvastatin 5-10mg/kg bid for 7 days and 14 days off treatment for 21 days Cohort 1: 7.5 mg/kg bid for 7 days 14 days off Cohort 2: 10 mg/kg bid for 7 days 14 days off Cohort 3: ( ) mg/kg bid for 7 days 14 days off (to be determined based on PK data of cohort 1 and 2) Q 3 weeks

DETAILED DESCRIPTION:
This is a Phase 1, open-label, single center, dose escalation study to evaluate the safety, tolerability and pharmacokinetics of high dose simvastatin in patients with GI cancers. Three dose levels will be evaluated. Simvastatin will be given at escalating dose of 7.5mg/kg bid, 10mg/kg bid and ( ) mg/kg bid for 7 days and off treatment for 14 days (Final dose will be determined based on PK data of cohort 1 and 2). The treatment will be repeated every 3 weeks. The cohort size of at least 3 and up to 6 patients ('rolling six design') will be employed to improve the rate of accrual of patients to cohorts close to the presumed therapeutic dose by reducing the need for late replacement of patients who become non-evaluable during the DLT assessment period, whilst not compromising collection of safety data. The total number of patients will depend upon the number of dose adjustments necessary. And intra-patient dose escalation is not allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 20 years of age on day of signing informed consent
3. Have histologically or cytologically confirmed diagnosis of colorectal cancer or gastric cancer
4. For colorectal cancer, patients who progressed after 5FU or capecitabine, irinotecan,oxaliplatin, bevacizumab and cetuximab treatment (cetuximab is only for KRAS/NRAS wild type)
5. For gastric cancer, patients who progressed after second line chemotherapy.
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Have evaluable disease based on RECIST v1.1 as determined by investigator.
8. Be willing to provide blood sample for PK analysis.
9. Ability to swallow and retain oral medication.
10. Demonstrate adequate organ function

Exclusion Criteria:

1. Prior history of statins within 12 months from the date of study entry
2. Patients with massive ascites or disseminated bone metastases
3. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
5. Has an active infection requiring systemic therapy.
6. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
7. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
8. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
9. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
10. Patients with CPK > ULN at baseline

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2018-01-04 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose | 12months
  maximum tolerated dose

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea